CLINICAL TRIAL: NCT01253122
Title: Comparative Bioavailability of TRx0037 and TRx0014 in Healthy Elderly Volunteers
Brief Title: Comparative Bioavailability in Healthy Elderly Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TauRx Therapeutics Ltd (Industry)
Collaborators: Quotient Clinical (Other)
Responsible Party: Professor Claude M. Wischik, Chairman, TauRx Therapeutics Ltd
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: TRx-037-002
Record Dates: First submitted 2010-12-02; First posted 2010-12-03 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-12

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TRx0037 (Experimental)
  Interventions: Drug: TRx0037
- TRx0014 (Active Comparator)
  Interventions: Drug: TRx0037

INTERVENTIONS:
Drug: TRx0037

SUMMARY:
A randomised four way crossover design in which each subject will receive two dose levels of TRx-0037 and two doses of TRx-0014 over approximately a four week period in randomised order.

ELIGIBILITY:
Inclusion Criteria:

* Male and female 55 and over
* No clinically important abnormal physical finding
* No clinically significant lab results
* Normal ECG, Normal BP and HR,BMI between 19 and 32
* Weight 50 to 100 kg, Able to communicate
* Provide written informed consent
* Non smokers
* Males to use contraception
* Females to be surgically sterile or post menopausal

Exclusion Criteria:

* Administration of any IMP other than study drug within 12 weeks before entry
* Use of any prescribed meds, St John's wort, over the counter meds as described in the protocol
* Surgical or medical condition that might interfere with IMP
* History of drug or alcohol abuse
* Clinically significant allergy requiring treatment
* Loss of greater than 400ml of blood within 12 weeks.
* Serious adverse reaction or hypersensitivity to any drug
* Prescence of Hep B, Hep c or HIV-1 or HIV-2 at screening
* Presence of G6PD at screening
* History of methaemoglobinaemia
* Partner who is pregnant of lactating
* Positive Pregnancy test

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-02; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Relative bioavailability
  Investigate the relative bioavailability of TRx0037 and TRx0014 at two molar equivalent doses in healthy elderly male and female (post-menopausal/non-childbearing) subjects

SECONDARY OUTCOMES:
Safety, tolerability and pharmacokinetics
  Safety, tolerability and pharmacokinetic (PK) evaluations of the two dose levels of TRx0037 and TRx0014.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Dr Mair, MBChB, Principal Investigator — Quotient Clinical